CLINICAL TRIAL: NCT00706641
Title: A Pilot Study of Neoadjuvant Dasatinib Followed by Radical Cystectomy for Transitional Cell Carcinoma of the Bladder
Brief Title: Neoadjuvant Dasatinib and Radical Cystectomy for Transitional Cell Carcinoma of the Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GU07-122
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Results first posted 2016-01-15 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2015-12

CONDITIONS: Transitional Cell Carcinoma of the Bladder
MeSH Terms: interventions — Dasatinib; Cystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental: Neoadjuvant Dasatinib + Radical Cystectomy (Experimental): Dasatinib 100 mg PO qd x 4 weeks followed by radical cystectomy 8-24 hours post last administered dasatinib dose
  Interventions: Drug: Dasatinib; Procedure: Radical Cystectomy

INTERVENTIONS:
Drug: Dasatinib — Dasatinib 100 mg administered orally once daily for 4 weeks duration (+/- 1 week)
Procedure: Radical Cystectomy — Radical cystectomy should be performed no sooner than 8 hours but preferably within 24 hours of the last administered Dasatinib dose. All attempts should be made for the patient to have their surgery after 8 hours but within 24 hours of their last dose of dasatinib. If surgery delay is imperative, dasatinib therapy should continue until at least 24 hours before planned surgery.

SUMMARY:
This pilot study is designed to determine feasibility and safety of treatment with dasatinib administered orally once daily for 4 weeks duration prior to radical cystectomy for urothelial carcinoma of the bladder.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

This is a pilot study designed to determine the safety and feasibility of treatment with dasatinib 100 mg administered orally once daily for 4 weeks duration prior to radical cystectomy for patients with muscle-invasive transitional cell carcinoma of the bladder ineligible for and/or willing to forgo neoadjuvant cisplatin-based combination chemotherapy. If surgery delay is imperative, dasatinib therapy should continue until at least 24 hours before planned surgery.

ECOG Performance Status 0-1

Life Expectancy: Not specified

Hematopoietic:

* Absolute Neutrophil Count (ANC) > 1.5 K/mm3
* Platelets > 100 K/mm3
* INR < 1.2

Hepatic:

* Total bilirubin < 2.0 X Upper Limit of Normal (ULN)
* Aspartate aminotransferase (AST) ≤ 2.5 X ULN.
* Alanine aminotransferase (ALT ) ≤ 2.5 X ULN

Renal:

* Serum creatinine < 2 X ULN

Cardiovascular:

* No uncontrolled angina, congestive heart failure or MI within 6 months prior to registration on study.
* No diagnosed congenital long QT syndrome (a congenital disorder characterized by a prolongation of the QT interval on ECG and a propensity to ventricular tachyarrhythmias, which may lead to syncope, cardiac arrest, or sudden death).
* No history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de Pointes).
* No prolonged QTc interval on pre-entry electrocardiogram (> 450 msec), obtained within 28 days prior to being registered on study.

ELIGIBILITY:
Inclusion Criteria:

* Histological proof of muscle-invasive transitional cell carcinoma of the bladder (stage II-IVa) with no evidence of metastatic disease (focal squamous and/or adenocarcinoma differentiation defined as ≤ 10% of tumor volume allowed, sarcomatoid and small-cell components not allowed). Patient with any degree of fixation of the pelvic sidewall are not eligible.
* Patients must be willing to undergo a Cystoscopy, prior to registration on study if tumor block is not available.
* Eligible for radical cystectomy as per the attending urologist.
* All patients must be willing to forego neoadjuvant cisplatin-based combination chemotherapy and understand it is an option post-surgery or must be deemed ineligible for cisplatin-based combination chemotherapy by the attending medical oncologist.
* Prior radiation therapy is allowed provided that no radiation therapy was administered to the urinary bladder.
* Written informed consent and HIPAA authorization for release of personal health information.
* Age > 18 years at the time of consent.
* Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time consent is signed until 4 weeks after treatment discontinuation.
* Females of childbearing potential must have a negative pregnancy test within 7 days prior to being registered for protocol therapy.
* Females must not be breastfeeding.
* Ability to take oral medication (dasatinib must be swallowed whole).

Exclusion Criteria:

* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, Gleason < grade 7 prostate cancers, or other cancer for which the patient has been disease-free for at least 5 years.
* No treatment with any investigational agent within 30 days prior to being registered for protocol therapy.
* No prior systemic chemotherapy for transitional cell carcinoma of the bladder( prior intravesical therapy is allowed). Any other prior chemotherapy must have been completed > 5 years prior to initiation of therapy.
* Following concomitant medications must be discontinued 7 days prior to registration on study and for the duration of dasatinib therapy: Bisphosphonates - due to risk of hypocalcemia; Drugs that are generally accepted to have a risk of causing Torsades de Pointes; any prohibited CYP3A4 inhibitors/inducers/substrates; Anti-coagulation and/or anti-platelet therapies to avoid potential bleeding risks.
* No clinically significant infections as judged by the treating investigator.
* No pleural or pericardial effusion of any grade.
* history of diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
* No history of diagnosed acquired bleeding disorder (e.g., acquired anti-factor VIII antibodies) within one year prior to registration on protocol therapy.
* No history of ongoing or recent (within <3 months prior to registration on protocol therapy) significant gastrointestinal bleeding.
* No known history of hypokalemia that cannot be corrected prior to registration on protocol therapy.
* No known history of hypomagnesemia that cannot be corrected prior to registration on protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noah Hahn, M.D., Study Chair — Hoosier Oncology Group, Inc.
Locations (3):
- United States (3):
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Baylor College of Medicine, Houston, Texas
  - Virginia Oncology Associates, Norfolk, Virginia

REFERENCES:
- [Background] Hahn NM, Knudsen BS, Daneshmand S, Koch MO, Bihrle R, Foster RS, Gardner TA, Cheng L, Liu Z, Breen T, Fleming MT, Lance R, Corless CL, Alva AS, Shen SS, Huang F, Gertych A, Gallick GE, Mallick J, Ryan C, Galsky MD, Lerner SP, Posadas EM, Sonpavde G. Neoadjuvant dasatinib for muscle-invasive bladder cancer with tissue analysis of biologic activity. Urol Oncol. 2016 Jan;34(1):4.e11-7. doi: 10.1016/j.urolonc.2015.08.005. Epub 2015 Sep 9. PMID 26362343
- See also: Hoosier Oncology Group Home Page — http://www.hoosieroncologygroup.org

RESULTS

PARTICIPANT FLOW:
Period: Dasatinib Administration
Arm/Group | Experimental: Neoadjuvant Dasatinib + Radical Cystectomy
Started | 25
Toxicity Evaluation | 24
Completed | 23
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Ineligible after start of therapy | 1
Period: Radical Cystectomy
Arm/Group | Experimental: Neoadjuvant Dasatinib + Radical Cystectomy
Started | 23
Completed | 22
Not Completed | 1
Not completed — Deemed unresectable upon exploration | 1

BASELINE CHARACTERISTICS:
Population: All subjects who started treatment on dastanib were included for age, gender, and ECOG PS characteristics. One patient was removed from the study because they were found to be ineligible based on histology after they started treatment and thus were not included in the T-Stage characteristics.
Arm/Group | Experimental: Neoadjuvant Dasatinib + Radical Cystectomy
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 62 [47 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 20
ECOG PS [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction and 5=Dead
  participants
    ECOG PS 0 | 19
    ECOG PS 1 | 6
T-Stage at Study Entry [Number; unit: participants] — Tumor Node Metastasis (TNM) Staging. This system classifies tumors by size and extent of the primary tumor (T), involvement of regional lymph nodes (N), and the presence or absence of distant metastases (M)
  T0=No evidence of primary tumor, Tis=Carcinoma in situ, and T1, T2, T3, T4=Increasing size and/or local extension of the primary tumor, TX=Not assessed N0=No Regional lymph node metastases, N1, N2, N3=Increasing number or extent of regional lymph node involvement, NX=not assessed M0=No distant metastases, M1=Distant metastases present
  participants
    T2 | 17
    T3 | 7
    T4a | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility
Description: Feasibility for this trial is defined as at least 60% (>=14 of 23) of patients completing study therapy in the absence of Dose Limiting Toxicity (DLT)
Time Frame: From enrollment to completion of radical cystectomy
Population: All patients who completed dasatinib
Measure: Number; unit: participants
Arm/Group | Experimental: Neoadjuvant Dasatinib + Radical Cystectomy
Number analyzed (Participants) | 23
participants
  DLT | 8
  Absence of DLT | 15

2. Secondary Outcome: Grade 3/4 Toxicities
Description: Report grade 3/4 toxicities during treatment with dasatinib prior to radical cystectomy in patients with muscle invasive transitional cell carcinoma of the bladder.
Time Frame: Time of consent through 30 days after treatment discontinuation
Population: 24 patients received treatment, 1 patient ineligible due to small cell histology after starting dasatinib treatment and was not evaluable.
Measure: Number; unit: percentage of particpants
Arm/Group | Experimental: Neoadjuvant Dasatinib + Radical Cystectomy
Number analyzed (Participants) | 24
percentage of particpants
  Anemia | 4
  Fatigue | 8
  Diarrhea | 4
  Nausea | 4
  Anorexia | 4
  Abdominal Pain | 4
  Dyspnea | 8
  Hematuria | 4
  Superventricular and Nodal Arrythmia | 4
  Enteric Fistula | 8
  Deep Vein Thrombosis \ Pulmonary Embolism | 8

3. Secondary Outcome: Reduced pSFK Expression
Description: pSFK levels were analyzed pre and post treatment
Time Frame: Baseline to post dasatinib therapy
Population: Sufficient tumor suitable for Immuno-Histochemistry (IHC) analysis was available from 20 patients
Measure: Number; unit: participants
Arm/Group | Experimental: Neoadjuvant Dasatinib + Radical Cystectomy
Number analyzed (Participants) | 20
participants | 16
Statistical Analysis 1: Comparison: Experimental: Neoadjuvant Dasatinib + Radical Cystectomy; Tumor samples from 20 patients were analyzed for expression of pSFK. A paired t-Test was used to calculate the significance of the difference in expression levels before and after treatment; Test type: Superiority or Other; p = 0.003, paired t-test

4. Secondary Outcome: Pathologic Complete Response (pCR) Rate
Description: Pathologic complete response (pCR) rate is defined as no residual evidence of muscle-invasive disease at cystectomy (< pT0).
Time Frame: 24 months
Population: 23 participants completed treatment and underwent radical cystectomy.
Measure: Number; unit: participants
Arm/Group | Experimental: Neoadjuvant Dasatinib + Radical Cystectomy
Number analyzed (Participants) | 23
participants | 0

5. Secondary Outcome: Post-Cystectomy Pathologic Stage
Description: Tumor Node Metastasis (TNM) Staging. This system classifies tumors by size and extent of the primary tumor (T), involvement of regional lymph nodes (N), and the presence or absence of distant metastases (M) T0=No evidence of primary tumor, Tis=Carcinoma in situ, and T1, T2, T3, T4=Increasing size and/or local extension of the primary tumor, TX=Not assessed N0=No Regional lymph node metastases, N1, N2, N3=Increasing number or extent of regional lymph node involvement, NX=not assessed M0=No distant metastases, M1=Distant metastases present
Time Frame: Staged Post-Cystectomy and dasatinib treatment
Measure: Number (95% Confidence Interval); unit: percentage of particpants
Arm/Group | Experimental: Neoadjuvant Dasatinib + Radical Cystectomy
Number analyzed (Participants) | 23
percentage of particpants
  T1\Tis | 23 [10 to 44]
  T2 | 27 [13 to 48]
  T3 | 41 [23 to 61]
  T4 | 9 [1 to 29]
  Unresectable | 5 [0 to 24]

6. Secondary Outcome: Reduced Ki-67 Expression
Description: Ki-67 levels were analyzed pre and post treatment
Time Frame: Baseline to post dasatinib therapy
Population: Sufficient tumor suitable for Immuno-Histochemistry (IHC) analysis was available from 20 patients
Measure: Number; unit: participants
Arm/Group | Experimental: Neoadjuvant Dasatinib + Radical Cystectomy
Number analyzed (Participants) | 20
participants | 4
Statistical Analysis 1: Comparison: Experimental: Neoadjuvant Dasatinib + Radical Cystectomy; Test type: Superiority or Other; p = 0.20, paired t-test

7. Secondary Outcome: Increase in Cas3 Expression
Description: Cas3 levels were analyzed pre and post treatment
Time Frame: Baseline to post dasatinib therapy
Population: Sufficient tumor suitable for Immuno-Histochemistry (IHC) analysis was available from 20 patients
Measure: Number; unit: participants
Arm/Group | Experimental: Neoadjuvant Dasatinib + Radical Cystectomy
Number analyzed (Participants) | 20
participants | 3
Statistical Analysis 1: Comparison: Experimental: Neoadjuvant Dasatinib + Radical Cystectomy; Test type: Superiority or Other; p = 0.42, paired t-test

ADVERSE EVENTS:
Time Frame: Duration of Study
Arm/Group | Experimental: Neoadjuvant Dasatinib + Radical Cystectomy
Serious Adverse Events (participants affected / at risk) | 4/25
Other Adverse Events (participants affected / at risk) | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Neoadjuvant Dasatinib + Radical Cystectomy (N=25)
ESOPHAGITIS (Gastrointestinal disorders) | 1 (1)
FISTULA, GI / ANUS (Gastrointestinal disorders) | 1 (1)
HEMORRHAGE, GI / PERITONEAL CAVITY (Gastrointestinal disorders) | 1 (1)
HYPERTENSION (Cardiac disorders) | 1 (1)
HYPOTENSION (Cardiac disorders) | 1 (1)
LEAK (INCLUDING ANASTOMOTIC), GI / SMALL BOWEL (Gastrointestinal disorders) | 1 (1)
PALPITATIONS (Cardiac disorders) | 1 (1)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA / ATRIAL FLUTTER (Cardiac disorders) | 1 (1)
THROMBOSIS/EMBOLISM (VASCULAR ACCESS-RELATED) (Vascular disorders) | 1 (1)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 1 (1)
WOUND COMPLICATION, NON-INFECTIOUS (Skin and subcutaneous tissue disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Neoadjuvant Dasatinib + Radical Cystectomy (N=25)
ALBUMIN, SERUM-LOW (HYPOALBUMINEMIA) (Investigations) | 2 (4)
ALKALINE PHOSPHATASE (Investigations) | 1 (1)
ALLERGIC RHINITIS (INCLUDING SNEEZING, NASAL STUFFINESS, POSTNASAL DRIP) (Immune system disorders) | 2 (2)
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 1 (1)
ANOREXIA (Gastrointestinal disorders) | 12 (15)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 1 (1)
ATAXIA (INCOORDINATION) (Nervous system disorders) | 2 (2)
BICARBONATE, SERUM-LOW (Investigations) | 2 (2)
BLADDER SPASMS (Renal and urinary disorders) | 4 (4)
CALCIUM, SERUM-LOW (HYPOCALCEMIA) (Investigations) | 1 (2)
CARDIAC GENERAL - OTHER (SPECIFY, __) (Cardiac disorders) | 2 (3)
CONSTIPATION (Gastrointestinal disorders) | 13 (17)
CONSTITUTIONAL SYMPTOMS - OTHER (SPECIFY, __) (General disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2)
CREATININE (Investigations) | 1 (1)
DERMATOLOGY/SKIN - OTHER (SPECIFY, __) (Skin and subcutaneous tissue disorders) | 3 (3)
DIARRHEA (Gastrointestinal disorders) | 13 (15)
DISTENSION/BLOATING, ABDOMINAL (Gastrointestinal disorders) | 2 (2)
DIZZINESS (Nervous system disorders) | 1 (1)
DRY MOUTH/SALIVARY GLAND (XEROSTOMIA) (Gastrointestinal disorders) | 2 (2)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 5 (8)
EDEMA: LIMB (Blood and lymphatic system disorders) | 2 (2)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 1 (1)
ESOPHAGITIS (Gastrointestinal disorders) | 1 (1)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 22 (32)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 2 (3)
FISTULA, GI / SMALL BOWEL NOS (Gastrointestinal disorders) | 1 (1)
FLUSHING (Skin and subcutaneous tissue disorders) | 2 (2)
GASTROINTESTINAL - OTHER (SPECIFY, __) (Gastrointestinal disorders) | 2 (2)
GLUCOSE, SERUM-HIGH (HYPERGLYCEMIA) (Investigations) | 4 (4)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 11 (15)
HEMOGLOBIN (Blood and lymphatic system disorders) | 6 (22)
HEMOGLOBINURIA (Investigations) | 2 (2)
HEMOLYSIS (E.G., IMMUNE HEMOLYTIC ANEMIA, DRUG-RELATED HEMOLYSIS) (Blood and lymphatic system disorders) | 1 (1)
HEMORRHAGE, GU / BLADDER (Gastrointestinal disorders) | 4 (7)
HEMORRHAGE, GU / URINARY NOS (Renal and urinary disorders) | 3 (5)
HEMORRHAGE/BLEEDING - OTHER (SPECIFY, __) (General disorders) | 1 (1)
HEMORRHAGE/BLEEDING ASSOCIATED WITH SURGERY, INTRA-OPERATIVE OR POSTOPERATIVE (Injury, poisoning and procedural complications) | 1 (1)
HEMORRHOIDS (Gastrointestinal disorders) | 1 (1)
HYPERTENSION (Cardiac disorders) | 4 (4)
INFECTION WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / BLADDER (URINARY) (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / BLADDER (URINARY) (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / URINARY TRACT NOS (Infections and infestations) | 3 (3)
INFECTION WITH UNKNOWN ANC / PERITONEAL CAVITY (Infections and infestations) | 1 (1)
INFECTION WITH UNKNOWN ANC / URINARY TRACT NOS (Infections and infestations) | 1 (1)
INFECTION WITH UNKNOWN ANC / VAGINA (Infections and infestations) | 1 (1)
INSOMNIA (General disorders) | 5 (6)
METABOLIC/LABORATORY - OTHER (SPECIFY, __) (Investigations) | 1 (1)
MOOD ALTERATION / ANXIETY (Psychiatric disorders) | 5 (5)
MOOD ALTERATION / DEPRESSION (Psychiatric disorders) | 4 (4)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) / ORAL CAVITY (Surgical and medical procedures) | 3 (3)
MUSCULOSKELETAL/SOFT TISSUE - OTHER (SPECIFY, __) (Musculoskeletal and connective tissue disorders) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 14 (26)
NEUROLOGY - OTHER (SPECIFY, __) (Nervous system disorders) | 1 (2)
NEUROPATHY: SENSORY (Nervous system disorders) | 3 (3)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1)
OBSTRUCTION, GU / BLADDER (Renal and urinary disorders) | 2 (2)
PAIN / ABDOMEN NOS (Gastrointestinal disorders) | 8 (10)
PAIN / BACK (General disorders) | 2 (2)
PAIN / BLADDER (Renal and urinary disorders) | 6 (7)
PAIN / BONE (Musculoskeletal and connective tissue disorders) | 1 (3)
PAIN / BUTTOCK (General disorders) | 1 (1)
PAIN / EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 2 (2)
PAIN / HEAD/HEADACHE (General disorders) | 5 (6)
PAIN / JOINT (Musculoskeletal and connective tissue disorders) | 3 (5)
PAIN / MUSCLE (Musculoskeletal and connective tissue disorders) | 1 (2)
PAIN / PAIN NOS (General disorders) | 2 (2)
PAIN / PELVIS (General disorders) | 2 (2)
PAIN / PENIS (Reproductive system and breast disorders) | 1 (1)
PAIN / RECTUM (Gastrointestinal disorders) | 1 (2)
PAIN / STOMACH (Gastrointestinal disorders) | 1 (1)
PAIN / TESTICLE (Reproductive system and breast disorders) | 1 (1)
PAIN / THROAT/PHARYNX/LARYNX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PAIN / TUMOR PAIN (General disorders) | 2 (3)
PAIN - OTHER (SPECIFY, __) (General disorders) | 7 (9)
PALPITATIONS (Cardiac disorders) | 2 (2)
PANCREATIC ENDOCRINE: GLUCOSE INTOLERANCE (Endocrine disorders) | 1 (1)
PLATELETS (Blood and lymphatic system disorders) | 1 (1)
POTASSIUM, SERUM-HIGH (HYPERKALEMIA) (Investigations) | 1 (1)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 6 (6)
PULMONARY/UPPER RESPIRATORY - OTHER (SPECIFY, __) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 2 (2)
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 3 (3)
RASH: HAND-FOOT SKIN REACTION (Skin and subcutaneous tissue disorders) | 2 (4)
RENAL FAILURE (Renal and urinary disorders) | 1 (1)
RENAL/GENITOURINARY - OTHER (SPECIFY, __) (Renal and urinary disorders) | 8 (12)
RIGORS/CHILLS (General disorders) | 2 (2)
SALIVARY GLAND CHANGES/SALIVA (Gastrointestinal disorders) | 1 (1)
SKIN BREAKDOWN/DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1 (1)
SODIUM, SERUM-LOW (HYPONATREMIA) (Investigations) | 1 (1)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA / ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA / SINUS TACHYCARDIA (Cardiac disorders) | 1 (1)
SWEATING (DIAPHORESIS) (General disorders) | 1 (1)
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 6 (7)
URINARY FREQUENCY/URGENCY (Renal and urinary disorders) | 7 (8)
URINARY RETENTION (INCLUDING NEUROGENIC BLADDER) (Renal and urinary disorders) | 1 (2)
URINE COLOR CHANGE (Renal and urinary disorders) | 1 (1)
URTICARIA (HIVES, WELTS, WHEALS) (Skin and subcutaneous tissue disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 7 (8)
WEIGHT GAIN (General disorders) | 1 (1)
WEIGHT LOSS (General disorders) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No